CLINICAL TRIAL: NCT04473469
Title: Previously Implanted Pudendal Nerve Stimulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Timothy Bruns, Associate Professor of Biomedical Engineering, Medical School, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00180124; OT2OD028191 (NIH)
Record Dates: First submitted 2020-07-13; First posted 2020-07-16 (Actual); Results first posted 2024-06-03 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Urinary Retention; Underactive Bladder
Keywords: Pudendal nerve mapping; Nerve stimulation
MeSH Terms: conditions — Urinary Retention; Urinary Bladder, Underactive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Cystometrogram (Experimental): The bladder will be filled to different volumes and electrical stimulation will be applied to the pudendal nerve via the implanted neurostimulator.
  Interventions: Device: Medtronic Interstim II Model 3058 Neurostimulator

INTERVENTIONS:
Device: Medtronic Interstim II Model 3058 Neurostimulator — Patients will undergo stimulation of the pudendal nerve. All stimulation parameters used will be within the normal hard-coded limits of the implantable pulse generator (IPG).

SUMMARY:
This study seeks to examine the response of the bladder to different pudendal nerve stimulation frequencies, by studying patients who have been previously-implanted with pudendal nerve neurostimulators.

DETAILED DESCRIPTION:
The pudendal nerve goes to the urethra, anus, and other areas of the pelvic floor. Electrical stimulation of this nerve can help with bladder, bowel, and sexual problems, and pelvic pain. Researchers do not fully understand how the nerve helps with these functions or how the anatomy is different between people. Successful stimulation of the pudendal nerve may help improve medical care for future patients with bladder problems, pelvic pain, bowel problems, and/or sexual problems.

ELIGIBILITY:
Inclusion Criteria:

* Previously received an implanted neurostimulator at the pudendal nerve
* Adult (18 or older), capable of providing own informed consent and communicating clearly with the research team
* Capable of speaking, reading, and understanding English, as all study questionnaires are standardized assessments only available in English.
* Capable of attending the experimental session

Exclusion Criteria:

* Pregnant or planning to become pregnant during study. If a woman of child- bearing potential wishes to participate in this study, they will be pre-screened with a test to detect pregnancy
* Currently has a urinary tract infection (UTI)
* Currently has or tested positive in the last 14 days for COVID-19, or is symptomatic for COVID-19
* Unwilling to allow de-identified data to be stored for future use or shared with other researchers

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-01-19 (Actual); Primary Completion 2023-05-02 (Actual); Study Completion 2023-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tim Bruns, Ph.D., Principal Investigator — University of Michigan; Priyanka Gupta, M.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
All de-identified IPD collected during the trial will be available.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Will be available twelve months following publication of study findings, or earlier.
Access Criteria: Anyone who wishes to access the data.
URL: https://sparc.science/data?type=dataset

REFERENCES:
- See also: Related Pudendal Nerve Stimulation Study — https://clinicaltrials.gov/ct2/show/NCT04236596

RESULTS

PARTICIPANT FLOW:
Groups:
- Cystometrogram: The bladder will be filled to different volumes and electrical stimulation will be applied to the pudendal nerve via the implanted neurostimulator. All stimulation parameters used will be within the normal hard-coded limits of the implantable pulse generator (IPG).
Period: Overall Study
Arm/Group | Cystometrogram
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cystometrogram
Number analyzed (Participants) | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.00 (14.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Evoked Bladder Contractions of at Least 20 Centimeters of Water (cmH2O) During Cystometrogram
Description: The results reflects the number of participants who experienced an evoked bladder contraction of at least 20 centimeters of water during stimulation of the pudendal nerve. Bladder contractions were evoked by applying nerve stimulation to the pudendal nerve through testing of the participant's implanted stimulator.
Time Frame: Visit 1, approximately 1 week after consent
Measure: Count of Participants; unit: Participants
Arm/Group | Cystometrogram
Number analyzed (Participants) | 5
Participants | 1

2. Secondary Outcome: Selective Stimulation of Pudendal Nerve Branches
Description: Selective stimulation of pudendal nerve branches for external urethral sphincter closure determined by comparing sensor recordings from distal pudendal nerve branches.
  The intention was to measure the effect of selective PNS, configured for selective external urethral sphincter stimulation on ULPP, but this selective stimulation for this nerve bundle, as described in the protocol, proved to not be feasible within the experimental sessions. Thus, no data was gathered.
Time Frame: 2 hours
Population: No participants had selective external urethral sphincter stimulation.
Arm/Group | Cystometrogram
Number analyzed (Participants) | 0

3. Secondary Outcome: Measurement of Effect of Selective Pudendal Nerve Stimulation (PNS) on Urethral Leak Point Pressure (ULPP)
Description: Measurement of effect of selective PNS on ULPP using PNS configured for external urethral sphincter selectivity.
  The intention was to measure the effect of selective PNS, configured for selective external urethral sphincter stimulation on ULPP, but this selective stimulation for this nerve bundle, as described in the protocol, proved to not be feasible within the experimental sessions. Thus, no data was gathered.
Time Frame: 2 hours
Population: No participants had selective external urethral sphincter stimulation.
Arm/Group | Cystometrogram
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 2 years, 3 months
Arm/Group | Cystometrogram
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2021-05-13): https://cdn.clinicaltrials.gov/large-docs/69/NCT04473469/Prot_000.pdf
  • Informed Consent Form (2023-03-05): https://cdn.clinicaltrials.gov/large-docs/69/NCT04473469/ICF_001.pdf